CLINICAL TRIAL: NCT02265588
Title: Reducing Symptoms of Depression and Anxiety in Adolescents With Inflammatory Bowel Disease in Order to Improve Quality of Life and the Clinical Course of Disease.
Brief Title: Healthy Approach to Physical and Psychological Problems in Youngsters With IBD (HAPPY-IBD).
Acronym: HAPPY-IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Reinier de Graaf Groep (Other); Albert Schweitzer Hospital (Other); Maasstad Hospital (Other); Haga Hospital (Other); Amphia Hospital (Other); Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.C. Escher, M.D., Ph.D, Prof. J.C. Escher, PhD, pediatric gastroenterologist, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL49147.078.14
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Bowel Disease (IBD); Ulcerative Colitis; Crohn's Disease; Anxiety; Depression
Keywords: Inflammatory bowel disease (IBD); Ulcerative colitis; Crohn's disease; Children; Adolescents; Anxiety; Depression; Cognitive behavioral therapy
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Anxiety Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Care as usual (No Intervention): Care as usual means receiving their regular medical care. This consists of the regular follow up visits at the gastroenterologist every 3 months.
- Cognitive Behavioral Therapy (Experimental): The intervention group receives regular medical care (care as usual) AND a cognitive behavioral therapy program called PASCET-PI. The therapy sessions will be performed by trained psychologist.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — A disease specific cognitive behavioral therapy program called PASCET-PI: The PASCET-PI model focuses on behavioral activation, cognitive restructuring and problem solving skills to change maladaptive behaviors, cognitions and coping strategies specific for IBD.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The presented study aims to reduce symptoms of depression and anxiety in adolescents with inflammatory bowel disease and increased symptoms of anxiety and depression by using the disease specific CBT program (PASCET-PI)in order to improve quality of life and to improve the clinical course of disease.

DETAILED DESCRIPTION:
1. Objective: The primary objective is to determine the efficacy of a disease specific cognitive behavioral therapy program in adolescents with IBD and increased symptoms of depression or anxiety on reducing symptoms of depression. Secondary objectives are to assess the effect of the CBT program on a) the clinical course of disease b) reducing symptoms of anxiety, and c) improving quality of life. We also aim to identify psychosocial and medical factors that predict or moderate the treatment response to CBT in adolescent with IBD.
2. Study design: The presented study is a multicenter randomized controlled trial (RCT), involving CBT versus care as usual (CAU), in young IBD patients with increased symptoms of self-reported depression or anxiety. There will be three follow-up moments, after 3 months or after the intervention and after 6 and 12 months.
3. Study population: Patients with IBD between 10-25 years and increased symptoms of depression or anxiety. We aim to include 100 patients, from which 50 patients will be randomized to the treatment condition (CBT and CAU) and 50 to the control group (CAU).
4. Intervention: A disease specific CBT program called PASCET-PI. The control group (CAU),will receive routine medical treatment (thus no additional psychosocial intervention) and will maintain their regular follow up visits at the gastroenterologist every 3 months.
5. Main study endpoints: Main outcome is reduction in symptoms of depression. Important secondary outcomes are the presence of clinical relapse and reduction of symptoms of anxiety. Other secondary outcomes, amongst others, are IBD activity scores, quality of life, psychosocial functioning, and adherence to medical treatment.
6. Nature and extent of the burden and risks associated with participation, benefit and group relatedness: At first, patients with IBD 10 -25 years of age will be screened for symptoms of depression and anxiety at T1. Patients with increased symptoms of self-reported depression or anxiety (scoring above an age and gender specific cut-off score for increased depressive or anxiety symptoms) are asked to participate in the RCT. For all included patients, 4 study visits will take place, these will be combined with regular checkup visits at the gastroenterologist. Questionnaires will need to be filled in online, taking approximately 1.5 hour per assessment for patients and approximately 1 hour per assessment for parents. At baseline a psychiatric assessment interview will be executed by an independent research clinical psychologist by phone (20 minutes). The same research clinical psychologist will conduct a short psychiatric assessment interview at the follow up visits 10minutes). At baseline and after 3 months blood samples (when patients undergo routine venous punctures) will be drawn.

For patients in the CBT group, 13 sessions (6 outpatient sessions, 7 by phone) and three parental sessions will take place in a hospital close to their home. Our study population consists of adolescents and young adults with IBD, as this is a specific group with high reported symptoms of depression and anxiety, therefore they will most likely benefit from the intervention. The risks associated with participation can be considered negligible and the burden minimal. For the time investment of completing the questionnaires participants will receive an incentive of 25 euro after the final assessment, which will be communicated at the start.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 10-25 years with diagnosed IBD
* Informed consent or assent by patients and (if necessary) parents

Exclusion Criteria:

* IBD patients with parental report of mental retardation
* IBD patients receiving psychopharmacological treatment (antidepressants or benzodiazepines) for depression or anxiety
* No mastery of the Dutch language
* IBD patients with diagnosed: Bipolar disorder, Schizophrenia/psychotic disorder, Autism spectrum disorders, Obsessive-compulsive disorder, Posttraumatic stress disorder/Acute stress disorder, or Substance use disorder
* Physician reported substance abuse (alcohol, drugs) in the past month
* Clinician reported Selective mutism
* IBD patients already participating in an (psychological of psychopharmacological) intervention study
* IBD patients who received 8 sessions of manualized cognitive behavioral therapy last year
* current psychological treatment

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Reduction in symptoms of depression (change from baseline) | 12 weeks and 52 weeks
  Measured by the Child Depression Inventory (CDI (10-17 years), Beck Depression Inventory (BDI; 18-25 years) and severity rating (interview): the Children's Depression Rating Scale (CDRS;10-12 years) and Adolescent Depression Rating Scale(ADRS;13-20 years), HAM-D: Hamilton Depression Rating Scale (21-25 year)

SECONDARY OUTCOMES:
Reduction in symptoms of anxiety (change from baseline) | 12 weeks and 52 weeks
  Measured by SCARED-NL: Screen for Anxiety Related Emotional Disorders (10-20 years), Hospital Anxiety and Depression Scale (HADS; 21-25 year) and severity rating by Pediatrix Anxiety Rating Scale (PARS) (10-20 years) ,Hamilton Anxiety Rating (HAM-A)(21-25 year)
General Quality of Life | 12 weeks and 52 weeks
  Assessed by the Child Health Related Quality of Life (TACQOL) (10-15 years) Adult Health Related Quality of Life (TAAQOL, 16-25 years)
Social Skills | 12 weeks
  Assessed by Social Skills Rating System (SSRS) (10-20years) Novotni SSC: Social Skills Checklist (21-25 year)
Social competence | 12 weeks
  Assessed by Youth Self Report (YSR) / Adult Self Report (ASR)
Disease specific quality of life | 12 weeks and 52 weeks
  Assessed by the IMPACT-III-NL (10-20years) IBDQ: Inflammatory Bowel Disease Questionnaire (21-25 year)
Disease Activity | 52 weeks
  Assessed by the Pediatric Ulcerative Colitis Activity Index (PUCAI) (10-20 years) Pediatric Crohn's Disease Activity Index (PCDAI) (10-20 years) CDAI: Crohn's Disease Activity Index (21-25 years) Partial Mayo Score (21-25 years) Physician Global Assessment (PGA)
Clinical relapse (number of flares) | 52 weeks
  10-20 Years: Relapse for CD is defined as PCDAI>30 or an increase of>15 points and intensification of medical treatment.
  Relapse for UC is defined as PUCAI > 34 or an increase of ≥20 points for UC and intensification of medical treatment.
  21-25 years: Partial Mayo score of 3 or higher with intensification of medical treatment Or CDAI≥ 150 and an increase in baseline CDAI score of ≥ 70 points and intensification of medical treatment
Maintaining remission | 52 weeks
  Remission is defined as PCDAI < 10 for CD and PUCAI < 10 for UC. CDAI < 150 and Mayo score ≤2 with no individual subscore > 1
Medication Usage (change from baseline) | 52 weeks
  Type and dosage of medication
Necessity of surgical intervention | 52 weeks
  Description of type and extent of surgical intervention
Adherence to therapy (change from baseline) | 52 weeks
  Assessed by the Morisky Medical Adherence Scale (MASS-8)
Health care utilization (change from baseline) | 52 weeks
  Assessed by standardized items derived from the questionnaires and Report of the treating physician.
Inflammatory markers | baseline and 12, 24 and 52 weeks
  Inflammatory markers will be measured at all time points (baseline and after 3,6,12 months) Inflammatory markers like BSE, CRP, faecal calprotectin

OTHER OUTCOMES:
Disease perception (change from baseline) | 12 weeks
  Assesses by the Brief Illness Perceptions Questionnaire (B-IPQ)
Cognitive coping styles (change from baseline) | 12 weeks
  Assesses by the Cognitive Emotion Regulation Questionnaire (CERQ)
Quality of sleep (change from baseline) | 12 weeks
  Assesses by the Sleep Self-Report (SSR) (10-20 years) PSQI: Pittsburgh Sleep Quality Index (21-25 year)
Demographic factors | 12 weeks
  Assesses by the Rotterdam's quality of life interview
Parental anxiety and depression | 12 weeks
  Assesses by the Depression, Anxiety and Stress Scale (DASS-21)
Life Events | 12 weeks
  Assesses by the Life events questionnaire from CERQ
Family Functioning (change from baseline) | 12 weeks
  Assesses by the Family Assessment Device (FAD)
Disease phenotypes | 52 weeks
  Assessed by the Paris Classification
Treatment Strategy | 52 weeks
  The treatment strategy, type and dosage of medication will be extracted from the medical file and report of the treating physician.
White blood cell RNA expression profiles (change from baseline) | 12 weeks
  Assessing immune status is done by analyzing gene expression profiles in peripheral blood leukocytes. This will be performed
Immunological activity in peripheral blood mononuclear cells (PBMC) | 12 weeks
  A blood sample will be taken in all patients included within the Erasmus MC for determination of responsiveness of peripheral blood lymphocytes before and directly after the intervention
Irritable bowel syndrome -like symptoms | 12 months
  Assessed by the ROME III diagnostic criteria for IBS in pediatric IBD patients

CONTACTS AND LOCATIONS:
Overall Officials: Johanna C. Escher, PhD, MD, Study Chair — Erasmus Medical Centre
Locations (1):
- Erasmus Medical Center, Rotterdam, Nederland, Netherlands

REFERENCES:
- [Background] Szigethy E, Kenney E, Carpenter J, Hardy DM, Fairclough D, Bousvaros A, Keljo D, Weisz J, Beardslee WR, Noll R, DeMASO DR. Cognitive-behavioral therapy for adolescents with inflammatory bowel disease and subsyndromal depression. J Am Acad Child Adolesc Psychiatry. 2007 Oct;46(10):1290-1298. doi: 10.1097/chi.0b013e3180f6341f. PMID 17885570
- [Background] Thompson RD, Craig A, Crawford EA, Fairclough D, Gonzalez-Heydrich J, Bousvaros A, Noll RB, DeMaso DR, Szigethy E. Longitudinal results of cognitive behavioral treatment for youths with inflammatory bowel disease and depressive symptoms. J Clin Psychol Med Settings. 2012 Sep;19(3):329-37. doi: 10.1007/s10880-012-9301-8. PMID 22699797
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Stapersma L, van den Brink G, van der Ende J, Szigethy EM, Groeneweg M, de Bruijne FH, Hillegers MHJ, Escher JC, Utens EMWJ. Psychological Outcomes of a Cognitive Behavioral Therapy for Youth with Inflammatory Bowel Disease: Results of the HAPPY-IBD Randomized Controlled Trial at 6- and 12-Month Follow-Up. J Clin Psychol Med Settings. 2020 Sep;27(3):490-506. doi: 10.1007/s10880-019-09649-9. PMID 31506853
- [Derived] Stapersma L, van den Brink G, van der Ende J, Szigethy EM, Beukers R, Korpershoek TA, Theuns-Valks SDM, Hillegers MHJ, Escher JC, Utens EMWJ. Effectiveness of Disease-Specific Cognitive Behavioral Therapy on Anxiety, Depression, and Quality of Life in Youth With Inflammatory Bowel Disease: A Randomized Controlled Trial. J Pediatr Psychol. 2018 Oct 1;43(9):967-980. doi: 10.1093/jpepsy/jsy029. PMID 29850915
- [Derived] van den Brink G, Stapersma L, El Marroun H, Henrichs J, Szigethy EM, Utens EM, Escher JC. Effectiveness of disease-specific cognitive-behavioural therapy on depression, anxiety, quality of life and the clinical course of disease in adolescents with inflammatory bowel disease: study protocol of a multicentre randomised controlled trial (HAPPY-IBD). BMJ Open Gastroenterol. 2016 Mar 2;3(1):e000071. doi: 10.1136/bmjgast-2015-000071. eCollection 2016. PMID 26966551